CLINICAL TRIAL: NCT04380337
Title: Phase II Trial of Organ Preservation Program Using Short-Course Radiation and FOLFOXIRI for Rectal Cancer (SHORT-FOX)
Brief Title: Organ Preservation Program Using Short-Course Radiation & FOLFOXIRI in Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Erqi Liu Pollom, Associate Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-56027; IRB-56027 (Other: Stanford IRB); COR0019 (Other: OnCore)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Folfox protocol; XELOX; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation/FOLFOXIRI (Experimental): Treatment will comprise 6 daily fractions of radiotherapy at 5 Gy per fraction followed by 4 months of FOLFOXIRI. Patients who have performance status or conditions that may preclude use of FOLFOXIRI may be treated with FOLFOX or XELOX. Those who achieve a clinical complete response will be considered for organ preservation approach. All other patients will receive standard of care total mesorectal excision (TME).
  Interventions: Drug: FOLFOXIRI; Drug: FOLFOX regimen; Drug: XELOX; Radiation: IMRT

INTERVENTIONS:
Drug: FOLFOXIRI — Chemotherapy regimen of Oxaliplatin 85mg/m2 , Leucovorin 400 mg/m2 , Irinotecan 165mg/m2 , 5-Fluorouracil
Drug: FOLFOX regimen — Chemotherapy regimen of Oxaliplatin 85mg/m2, Leucovorin 400 mg/m2, 5-Fluorouracil 2400mg/m2
Drug: XELOX — Chemotherapy regimen of Oxaliplatin 130 mg/m2, Capecitabine 1000mg/m2
Radiation: IMRT — Radiotherapy (5 Gy x 5 fractions) with an additional boost fraction (5 Gy x 1 fraction) delivered sequentially
  Other Names: Intensity-modulated radiotherapy (IMRT)

SUMMARY:
The purpose of the research is to evaluate whether both chemotherapy and radiotherapy can lead to higher rates of clinical complete response leading to organ preservation in human subjects with cancer. The objective is to learn if this treatment approach may safely be used as an alternative to the standard treatment for rectal cancer and to know the quality-of-life in these patients.

DETAILED DESCRIPTION:
Primary Objective: To assess clinical complete response of an organ preservation approach using short course radiation followed by intensified chemotherapy.

Secondary Objective: To assess safety in all enrolled patients, local regrowth rate and other cancer specific outcomes (metastasis-free survival, colostomy-free survival and overall survival), longitudinal health-related quality of life of this organ preservation approach

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma of rectum requiring total mesorectal excision as deemed by multidisciplinary evaluation
* 2.At least 18 years of age
* 3.For women of childbearing potential or who are not postmenopausal (see Appendix B for Definition of Menopausal Status), a negative urine or serum pregnancy test must be done. Also, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for up to 4 weeks following the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* 4.ECOG 0, 1, or 2
* 5.Ability to understand and the willingness to personally sign the written IRB approved informed consent document.
* 6.Patients must have acceptable organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >1,500/uL
  * Hg > 8.0 g/dL; if blood transfusion is performed for achieving adequate hemoglobin level, the level should stay above goal for at least 1 week after transfusion
  * Platelets >100,000/uL
  * Total bilirubin <1.5X normal institutional limits
  * aspartate aminotransferase (AST) (SGOT) / alanine aminotransferase (ALT)(SGPT) < 3X upper limit of normal
  * Creatinine <1.5X upper limit of normal or creatinine clearance (CrCL)>50 by Cockcroft-Gault
* 7 Clinical stage >T2N0 or low T2N0 rectal cancer (AJCC, 8th ed.) including no metastases based on the following diagnostic workup:

  * General history and physical examination with DRE (if deemed appropriate by treating physician) within 45 days prior to enrollment
  * Sigmoidoscopy within 90 days prior to enrollment

The following imaging studies are required within 45 days prior to enrollment:

* CT chest/abdomen/pelvis
* MRI Pelvis

Exclusion Criteria:

* 1.Prior pelvic RT or chemotherapy for rectal cancer.
* 2.Upper T2N0 rectal cancers eligible for sphincter-preservation surgery
* 3.Use of other investigational agents.
* 4.Ongoing or active infections requiring systemic antibiotic treatment or uncontrolled intercurrent illness including but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* 5.Any concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix. Patients with any previous malignancy without evidence of disease for >3 years will be allowed to enter the trial.
* 6.Known hypersensitivity to 5-FU compounds.
* 7.Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study are excluded. (This applies to women who have experienced menarche and have not undergone successful surgical sterilization or are not postmenopausal).

Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, known HIV-positive patients with detectable viral loads and/or receiving combination anti-retroviral therapy are excluded from the study.

- 8.Primary unresectable rectal cancer (tumor invading adjacent organs and en bloc resection will not achieve negative margins).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erqi L Pollom, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown E, Fisher GA Jr, Shelton A, Chang DT, Pollom E. Advancing clinical trial equity through integration of telehealth and decentralized treatment. JNCI Cancer Spectr. 2024 Jul 1;8(4):pkae050. doi: 10.1093/jncics/pkae050. PMID 38902952

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 patients were enrolled, but 1 withdrew prior to treatment start and was thus "replaced". We had 37 patients initiate treatment on study and be evaluable for primary outcome.
Groups:
- Radiation/FOLFOXIRI: Treatment comprised of 6 daily fractions of radiotherapy at 5 Gy per fraction followed by 4 months of FOLFOXIRI.
Period: Overall Study
Arm/Group | Radiation/FOLFOXIRI
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Clinical Complete Response (cCR)
Description: Proportion of patients who achieve a clinical complete response following therapy, expressed as a number and proportion without dispersion.
Time Frame: 8 (+/-4 ) weeks following completion of RT and chemotherapy, an average of 9 months
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
Proportion of Participants | 0.24 [0.105 to 0.381]

2. Secondary Outcome: Number of Participants With Toxicity
Description: Toxicity defined as non-hematologic grade 4 adverse events using CTCAE v5 or higher toxicity at least possibly related to treatment, and assessed up to 3 months after completion of radiotherapy (RT) and chemotherapy.
Time Frame: 8 (+/- 4) weeks following completion of RT and chemotherapy, an average of 3 months
Measure: Number; unit: proportion of participants
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
proportion of participants | 0

3. Secondary Outcome: Local Regrowth Rate
Description: Local regrowth is defined as the presence of adenocarcinoma within the rectal wall or within the mesorectum confirmed by pathology, expressed as a percentage with its 95% confidence interval.
Time Frame: 22 (+/- 2) months following completion of RT and chemotherapy, an average of 24 months (2 years)
Population: All patients managed with an organ preservation approach.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 18
Percentage of participants | 50 [26 to 74]

4. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS defined as the time from the start date of RT to the date of the first documented progression or death due to any cause assessed up to 2 years after completion of chemotherapy. Patients will be censored at the last date of follow-up if lost to follow-up prior to two years, expressed as a median with interquartile range.
Time Frame: 22 (+/- 2) months following completion of RT and chemotherapy, an average of 24 months (2 years)
Population: All participants who initiated the RT and chemotherapy regimen (intent-to-treat population) were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
months | 22 [18 to 28]

5. Secondary Outcome: Colostomy-free Survival
Description: Colostomy-free survival defined as the time from the start date of RT to the date of colostomy or death due to any cause assessed up to 2 years after completion of chemotherapy, expressed as a median with interquartile range. Patients will be censored at the last date of follow-up if lost to follow-up prior to two years.
Time Frame: 22 (+/- 2) months following completion of RT and chemotherapy, an average of 24 months (2 years)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
months | 11 [8 to 18]

6. Secondary Outcome: Overall Survival (OS)
Description: OS defined as death from any cause from start date of RT until death, study completion, or loss to follow-up, whichever occurs first. This will be reported as median survival time with interquartile range.
Time Frame: 27 (+/- 4) months following completion of RT and chemotherapy, an average of 2.25 years
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Radiation/FOLFOXIRI
Number analyzed (Participants) | 37
months | 27 [19 to 31]

ADVERSE EVENTS:
Time Frame: 27 (+/- 4) months following completion of RT and chemotherapy, an average of 2.25 years
Arm/Group | Radiation/FOLFOXIRI
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 25/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation/FOLFOXIRI (N=37)
Lower GI Hemorrhage (Gastrointestinal disorders) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Vasovagal Reaction (Nervous system disorders) | 2 (2)
ALT Increase (Investigations) | 1 (1)
Catheter Related Infection (Infections and infestations) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
abcess (Injury, poisoning and procedural complications) | 1 (1) — pelvic abcess
Myelitis (Infections and infestations) | 1 (1)
Pelvic Infection (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
stoma (Injury, poisoning and procedural complications) | 1 (1) — prolapse of intestinal stoma
Thromboembolic Event (Vascular disorders) | 1 (1)
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Lymphocyte count decrease (Investigations) | 10 (11)
Rectal Pain (Gastrointestinal disorders) | 3 (5)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decrease (neutropenia) (Investigations) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 5 (5)
WBC decrease (Investigations) | 3 (3)
Anemia (Investigations) | 2 (2)
Rectal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation/FOLFOXIRI (N=37)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 19 (25)
ALKALINE PHOSPHATASE INCREASE (Investigations) | 26 (33)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17)
ANAL FISSURE (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 30 (42)
ANOREXIA (Metabolism and nutrition disorders) | 6 (8)
ANOSMIA (Nervous system disorders) | 3 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 14 (18)
BLOATING (Gastrointestinal disorders) | 6 (9)
BLOOD BILIRUBIN INCREASE (Investigations) | 1 (1)
BLURRED VISION (Eye disorders) | 4 (5)
General Disorders - other, body ache (General disorders) | 1 (1)
Gastrointestinal Disorders - other, anorectal spasm (Gastrointestinal disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
General Disorders - other, COLD LIKE SYMPTOMS (General disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (18)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (9)
CREATININE INCREASE (Investigations) | 2 (3)
CYSTIS NONINFECTIVE (Renal and urinary disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 26 (69)
DIZZINESS (Nervous system disorders) | 6 (7)
DRY EYE (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 5 (6)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 13 (21)
DYSPEPSIA (Gastrointestinal disorders) | 8 (14)
Dysphagia (Gastrointestinal disorders) | 2 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
DYSURIA (Renal and urinary disorders) | 7 (8)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
EYE DISORDERS-- OTHER PERIPHERAL VISION LOSS (Eye disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 33 (89)
FECAL INCONTINENCE (Gastrointestinal disorders) | 5 (5)
FEVER (General disorders) | 3 (5)
FLATULENCE (Gastrointestinal disorders) | 7 (8)
FLU-LIKE SYMPTOMS (General disorders) | 3 (3)
FLUSHING (Vascular disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (7)
GI DISORDER - DYSCHEZIA (Gastrointestinal disorders) | 1 (1)
GI DISORDER - FOOD SENSITIVITIES RESULTING IN DIARRHEA (Gastrointestinal disorders) | 1 (1)
GI DISORDERS - OTHER, TENESMUS (Gastrointestinal disorders) | 3 (6)
Headache (Nervous system disorders) | 9 (13)
HEMATURIA (Renal and urinary disorders) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders - OTHER, HEMOPYTSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 9 (18)
HOT FLASHES (Vascular disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 6 (8)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 6 (10)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 10 (15)
INJURY, POISIONING AND PROCEDURAL COMPLICATIONS - OTHER, INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1)
INSOMNIA (Psychiatric disorders) | 7 (8)
LOCALIZED EDEMA (FEET) (General disorders) | 1 (2)
Lymphocyte count decrease (Investigations) | 23 (36)
MALAISE (General disorders) | 2 (6)
MUCOSITIS ORAL (Gastrointestinal disorders) | 11 (15)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 9 (19)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 33 (115)
NERVOUS SYSTEM DISORDER - JAW CLAUDICATION (Nervous system disorders) | 5 (11)
Neutrophil count decrease (Investigations) | 5 (5)
INFECTIONS AND INFESTATIONS - OTHER, BLASTOCYSTIS HOMINIS AND ENTAMOEBA COLI CYSTS (Infections and infestations) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
Injury, Poisoning and Procedural Complications - other, OSTOMY LEAK (Injury, poisoning and procedural complications) | 1 (1)
Pain - Abdominal (Gastrointestinal disorders) | 16 (23)
Pain - ANAL (Gastrointestinal disorders) | 1 (1)
Pain - AT PORT SITE (General disorders) | 2 (2)
Pain - AT SURGICAL SITE (General disorders) | 4 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain - BILATERAL ARMS (General disorders) | 1 (1)
Pain - BONE (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain - EAR (Ear and labyrinth disorders) | 1 (1)
Pain - EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain - EYE (Eye disorders) | 1 (1)
Pain - FLANK (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - NECK (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - ORAL (Gastrointestinal disorders) | 1 (1)
Pain - PERIANAL (Reproductive system and breast disorders) | 1 (1)
Pain - Rectal (Gastrointestinal disorders) | 16 (21)
Pain - SCALP (Skin and subcutaneous tissue disorders) | 1 (1)
Pain - SHOULDER (General disorders) | 1 (1)
PAIN AT SURGICAL SITE (General disorders) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2)
PAPULOPUSTULAR RASH (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 34 (124)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 21 (32)
PHOTOPHOBIA (Eye disorders) | 2 (4)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decrease (Investigations) | 22 (29)
Reproductive System and Breast Disorders - Other, PRESSURE AT TESTICULAR AREA (Reproductive system and breast disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 2 (3)
Proctitis (Gastrointestinal disorders) | 23 (28)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4)
RECTAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 12 (13)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY MENSTRUAL SPOTTING (Reproductive system and breast disorders) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 1 (3)
Reproductive System and Breast Disorders - Other, LABIA DISCOMFORT (Reproductive system and breast disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER,TWO FEET ONE HAND SYNDROME (TFOHS) (Skin and subcutaneous tissue disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Gastrointestinal Disorders - other, STOOL URGENCY (Gastrointestinal disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
THRUSH (Infections and infestations) | 4 (8)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
TREMOR (Nervous system disorders) | 2 (2)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 7 (7)
URINARY INCONTINENCE (Renal and urinary disorders) | 4 (4)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
URINARY URGENCY (Renal and urinary disorders) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 17 (41)
WBC decrease (Investigations) | 19 (30)
WEIGHT GAIN (Investigations) | 1 (1)
WEIGHT LOSS (Investigations) | 14 (15)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT04380337/Prot_SAP_000.pdf